CLINICAL TRIAL: NCT01145898
Title: Trusopt and Cosopt; Ocular Perfusion Pressure and Blood Flow: New Long-term Prospective Data
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: Cosopt and OAG progression
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma
Keywords: Glaucoma; Cosopt; blood flow; progression
MeSH Terms: conditions — Glaucoma; Disease Progression | interventions — dorzolamide-timolol combination; Prostaglandins; Timolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma patients: Patients with Glaucoma
  Interventions: Drug: (Cosopt®, prostaglandin)

INTERVENTIONS:
Drug: (Cosopt®, prostaglandin) — We did NOT provide any intervention, we observed groups of patients already on these drugs as observers only.
  Other Names: Cosopt is a trade name drug which is a combination of dorzolamide and timolol.

SUMMARY:
To analyze Cosopt® in terms of its effects on ocular perfusion pressure and comprehensive ocular blood flow and in relation to visual field progression and optic nerve structural changes in an ongoing 3 year prospective study involving 120 patients with open angle glaucoma.

DETAILED DESCRIPTION:
To analyze Cosopt® in terms of its effects on ocular perfusion pressure and comprehensive ocular blood flow and in relation to visual field progression and optic nerve structural changes in an ongoing 3 year prospective study involving 120 patients with open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30 years or older.
2. Diagnosis: confirmed open-angle glaucoma in at least one eye:

   1. glaucomatous visual field loss on Humphrey 24-2 or 10-2 perimetry
   2. glaucomatous optic disc cupping
   3. agreement between two baseline exams for reliability
3. Best corrected visual acuity at least 20/60 in at least one eye.
4. Prior Humphrey visual fields demonstrate acceptable reliability standards.

Exclusion Criteria:

1. Extensive Humphrey visual field damage consisting of either a mean deviation (MD) < -15 decibels or a clinically determined threat to fixation in both hemifields.
2. Evidence of exfoliation or pigment dispersion.
3. History of acute angle-closure or a narrow, occludable anterior chamber angle by gonioscopy.
4. History of chronic or recurrent inflammatory eye diseases (e.g., scleritis, uveitis).
5. History or signs of intraocular trauma.
6. Severe or potentially progressive retinal disease such as retinal degeneration, diabetic retinopathy, and retinal detachment.
7. Any abnormality preventing reliable applanation tonometry.
8. Current use of any ophthalmic or systemic steroid which may interfere with this investigation.
9. Cataract surgery within the past year.
10. Resting pulse < 50 beats per minute.
11. Severe, unstable or uncontrolled cardiovascular, renal, or pulmonary disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Department of Ophthalmology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment over 6 months. Hospital and area eye clinics
Pre-assignment Details: observational study, patients were treated by their physician not by study personel, treatments/interventions were self-reported by the patients, treatment was not necessarily started at glaucoma diagnosis
Groups:
- Trusopt: Patients with glaucoma taking Trusopt or Cosopt alone or with prostaglandin for at least 6 months
- Prostaglandin Alone: Patients with glaucoma taking prostaglandin alone for at least 6 months
Period: 6-month Treatment
Arm/Group | Trusopt | Prostaglandin Alone
Started | 12 | 44
Completed | 12 | 44
Not Completed | 0 | 0
Period: 3-year Treatment
Arm/Group | Trusopt | Prostaglandin Alone
Started | 12 | 44
Completed | 9 | 28
Not Completed | 3 | 16
Not completed — medication change by treating physician | 3 | 16

BASELINE CHARACTERISTICS:
Population: glaucoma patients:There will be (as shown) differences in the number of subjects based upon the time of analysis due to patient loss, data of insufficient quality at visit, or change in the drug use during period of study (patient switched off treatment by their doctor) so the number of data points varies throughout the analysis by availability.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trusopt | Prostaglandin Alone | Total
Number analyzed (Participants) | 12 | 44 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 17 | 24
  >=65 years | 5 | 27 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.23 (6.78) | 65.25 (8.78) | 64.82 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 31 | 36
  Male | 7 | 13 | 20
Region of Enrollment [Number; unit: participants]
  United States | 12 | 44 | 56

OUTCOME MEASURES:

1. Primary Outcome: 6-month Change in Ophthalmic Artery (OA) Peak Systolic Velocity (PSV)
Description: Measurement of change in ocular blood flow - ophthalmic artery peak systolic velocity
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Groups:
- Trusopt: Patients taking trusopt or cosopt alone or with prostaglandin
- Prostaglandin Alone: Patients taking prostaglandin alone
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
cm/sec | 2.32 (1.20) | -.30 (1.17)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; There will be (as shown) differences in the number of subjects based upon the time of analysis due to patient loss, data of insufficient quality at visit, or change in the drug use during period of study (patient switched off treatment by their doctor) so the number of data points varies throughout the analysis by availability; Test type: Superiority or Other; p = .6261, ANCOVA

2. Primary Outcome: 6-month Change inOphthalmic Artery (OA) End Diastolic Velocity (EDV)
Description: Measurement of change in ocular blood flow - ophthalmic artery end diastolic velocity
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
cm/sec | .78 (.63) | -.03 (.39)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .6081, ANCOVA

3. Primary Outcome: 6-month Change in Ophthalmic Artery (OA) Vascular Resistance (RI)
Description: Measurement of change in ocular blood flow - ophthalmic artery resistance index, this is a measure of the amount of resistance to blood flow within the selected blood vessel.
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
unitless | -.011 (.020) | .002 (.008)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .1822, ANCOVA

4. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) Peak Systolic Velocity (PSV)
Description: Measurement of change in ocular blood flow - central retinal arteries peak systolic velocity
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
cm/sec | 0.24 (.34) | -.045 (.15)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .2383, ANCOVA

5. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) End Diastolic Velocity (EDV)
Description: Measurement of change in ocular blood flow - central retinal arteries end diastolic velocity
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
cm/sec | .18 (.16) | -.12 (.07)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .2383, ANCOVA

6. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) Vascular Resistance (RI)
Description: Measurement of change in ocular blood flow - central retinal arteries resistance index, this is a measure of the amount of resistance to blood flow within the selected blood vessel.
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
unitless | -.012 (.012) | .005 (.008)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .1564, ANCOVA

7. Primary Outcome: 6-month Change in Ocular Perfusion Pressures (OPP)
Description: Measurement of change in ocular perfusion pressure, the pressure of blood flow to the eye minus the pressure of within the eye.
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 12 | 44
mm Hg | -.30 (2.02) | -2.88 (1.06)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .2265, ANCOVA

8. Primary Outcome: 3-year Change in OA PSV
Description: Measurement of change in ocular blood flow - ophthalmic artery peak systolic velocity
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
cm/sec | -.62 (2.41) | .07 (1.25)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .4645, ANCOVA

9. Primary Outcome: 3-year Change in OA EDV
Description: Measurement of change in ocular blood flow - ophthalmic artery end diastolic velocity
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
cm/sec | -.58 (.58) | -.98 (.35)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .5998, ANCOVA

10. Primary Outcome: 3-year Change in OA RI
Description: Measurement of change in ocular blood flow - ophthalmic artery resistance index
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
unitless | .042 (.026) | .036 (.013)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .8119, ANCOVA

11. Primary Outcome: 3-year Change in CRA PSV
Description: Measurement of change in ocular blood flow - central retinal arteries peak systolic velocity
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
cm/sec | -.66 (.61) | .37 (.40)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .1319, ANCOVA

12. Primary Outcome: 3-year Change in CRA EDV
Description: Measurement of change in ocular blood flow - central retinal arteries end diastolic velocity
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
cm/sec | -.21 (.21) | .12 (.13)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .0199, ANCOVA

13. Primary Outcome: 3-year Change in CRA RI
Description: Measurement of change in ocular blood flow - central retinal arteries resistance index
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
unitless | .007 (.024) | .013 (.014)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .7597, ANCOVA

14. Primary Outcome: 3-year Change in OPP
Description: Measurement of change in ocular perfusion pressure
Time Frame: Baseline and 36 month visits
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Trusopt | Prostaglandin Alone
Number analyzed (Participants) | 9 | 27
mm Hg | -4.91 (2.74) | -1.43 (1.50)
Statistical Analysis 1: Comparison: Trusopt vs Prostaglandin Alone; Test type: Superiority or Other; p = .2528, ANCOVA

ADVERSE EVENTS:
Description: Adverse events were not assessed/collected as part of this study protocol.
Arm/Group | Glaucoma Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Small numbers of participants at various time-points limited the power of analysis in our estimation, as did patients who changed medications and therefore further limited analysis options at various time-points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No